CLINICAL TRIAL: NCT04779957
Title: Evaluation of the Safety of Use of Anti-IL6 Receptor Antibodies to Reduce Allo-sensitization Post Allograft Nephrectomy ; a Pilot Phase II Study.
Brief Title: Evaluation of the Safety of Use of Anti-IL6 Receptor Antibodies to Reduce Allo-sensitization Post Allograft Nephrectomy
Acronym: RAIPONS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/19/0511
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Kidney Transplantation; Graft Failure
Keywords: Kidney transplantation; allosensitization; graft nephrectomy; Donor-Specific Antibodies
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tocilizumab (Experimental): Evaluation of the use of Tocilizumab after allograft nephrectomy.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab will be administered at 8 mg/kg before or immediately after graft nephrectomy.

SUMMARY:
Graft nephrectomy is associated with massive allo-sensitization following this event. The occurrence of anti-HLA antibodies is a major barrier to perform a second kidney transplantation. Investigators propose here to evaluate in a phase II pilot study, the safety of the use of a single dose of Tocilizumab immediately before or after graft nephrectomy. The primary endpoint evaluated here is the occurrence of serious infectious complications following graft nephrectomy, with a treatment by Tocilizumab. Secondary endpoints evaluated here are - to evaluate all complications after graft nephrectomy, - and the Tocilizumab effectiveness to reduce anti-HLA antibodies at one year post nephrectomy.

DETAILED DESCRIPTION:
Background: graft nephrectomy is associated with massive allo-sensitization following this event The occurrence of anti-HLA antibodies is a major barrier to perform a second kidney transplantation. Moreover, a systemic inflammatory response syndrome can occur which could lead to serious patient's complications, in case of early graft thrombosis. To date, no treatment or strategy is available to reduce these risks, after graft nephrectomy. IL-6 is a key cytokine in inflammation, but also in the development of T and B cells activation. This treatment previously demonstrated a major role in the occurrence of allo-antibodies. Tocilizumab is a monoclonal antibody blocking IL6 receptor, previously used with success in kidney transplantation to reduce anti-HLA antibodies mediated rejection.

Objectives: Investigators hypothesize that Tocilizumab is useful to prevent allo-sensitization post graft nephrectomy. They propose here to evaluate in a phase II pilot study, the safety of the use of a single dose of Tocilizumab immediately before or after graft nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult recipients,
* affiliated to the social security
* requiring a graft nephrectomy, with a project to retransplantation

Exclusion Criteria:

* combined transplantations, PRA >20%.
* Patient under protective measures,
* Rituximab used for immunosuppression induction
* Previous transplants not removed,
* Active infectious complications at graft nephrectomy, need for immunosuppressive treatments after graft nephrectomy,
* Participation to another interventional studies using Rituximab, polyclonal antibodies, Eculizumab, or Tocilizumab.
* adults under guardianship or other legal protection, deprived of their liberty by judicial or administrative decision,
* pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
serious infectious complication | 1 year post graft nephrectomy
  serious infectious complication rate at 1 year post graft nephrectomy

SECONDARY OUTCOMES:
Complications after treatment | 1 year post graft nephrectomy
  Safety excluding serious infectious complications one year after nephrectomy, used by:
  * The occurrence of post-nephrectomy complications
  * The occurrence of death
  * The occurrence of hospitalizations
  * The occurrence of surgical complications
  * The occurrence of infectious complications (mild and moderate)
The effectiveness of the treatment | 1 year post graft nephrectomy
  The effectiveness of the treatment assessed by the rate of immunization after a post nephrectomy

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud DEL BELLO, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France